CLINICAL TRIAL: NCT02935075
Title: Optimization of Antiretroviral Therapy
Acronym: OAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Public Health Clinical Center (Other Government)
Collaborators: Yunnan Provincial Infectious Disease Hospital (Other); The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hongzhou Lu, Doctor, Shanghai Public Health Clinical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-M-1
Record Dates: First submitted 2016-10-14; First posted 2016-10-17 (Estimated); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir; Lamivudine; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduced dose (Experimental): Tenofovir 200mg +lamivudine 300mg +efavirenz 400mg PO q.d.
  Interventions: Drug: Tenofovir disoproxil fumarate; Drug: Lamivudine; Drug: Efavirenz
- Standard dose (Active Comparator): Tenofovir 300mg +lamivudine 300mg +efavirenz 600mg PO q.d.
  Interventions: Drug: Tenofovir disoproxil fumarate; Drug: Lamivudine; Drug: Efavirenz

INTERVENTIONS:
Drug: Tenofovir disoproxil fumarate — Oral daily
Drug: Lamivudine — Oral daily
Drug: Efavirenz — Oral daily

SUMMARY:
The combination antiretroviral therapy (cART) inhibit HIV replication effectively. However, synergy among these drugs has not been well considered. The dose of drugs used as monotherapy is the same as that used in combination therapy. Tenofovir+lamivudine+efavirenz is still the first line regimen of cART in developing countries. The side effects of these drugs are related to the concentration of drugs. Based on our previous data, we aim to evaluate whether reduce the dose of tenofovir and efavirenz could decreasing the incidence of the side effects while not scarifying their virological efficacy.

ELIGIBILITY:
Inclusion Criteria:

* HIV antibody positive
* Chinese nationality
* Naïve to antiretroviral therapy
* Willing to start antiretroviral therapy
* Provision of written informed consent

Exclusion Criteria:

* Pregnant, breastfeeding, or lactating
* Females try to get pregnant during the research period
* Subjects who allergic to any of the research drugs
* Subjects that taking other drugs that known to impact the absorption, distribution, metabolism and excretion of the research drugs
* Any serious or active medical or psychiatric illness which, in the opinion of the Investigator, would interfere with treatment, assessment, compliance with the protocol, or subject safety. This would include any active clinically significant renal, cardiac, pulmonary, vascular, or metabolic (thyroid disorders, adrenal disease) illness, or malignancy
* Medical or psychiatric condition or occupational responsibilities that may preclude compliance with the protocol
* Laboratory blood values:
* Haemoglobin <9.0 grams/decilitre (g/dL)
* Neutrophil count <1500/mm3
* Platelet count <75,000/mm3
* Aspartate aminotransferase or Alanine transaminase >3 times Upper Limit of Normal (ULN)
* Total bilirubin >3 times Upper Limit of Normal (ULN)
* Subjects with an estimated creatinine clearance of <90 mL/minute

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 184 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with HIV viral road < 50 copies/ml | 48 weeks
  calculate the percentage of patients who with HIV viral road <50 copies/ml every month in two groups

SECONDARY OUTCOMES:
Cell Differentiation 4 (CD4) T cell counts | 48 weeks

OTHER OUTCOMES:
The incidence of adverse events | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hongzhou Lu, Principal Investigator — Shanghai Public Health Clinical Center
Locations (3):
- China (3):
  - The Second Hospital of Nanjing, Nanjing, Jiangsu
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality
  - Yunnan AIDS care center, Kunming, Yunnan